CLINICAL TRIAL: NCT03022227
Title: Comparison of Remote Versus Standard On-site Care for Long Term Follow-up of Adult Cochlear Implant Users: a Prospective Controlled Feasibility Study
Brief Title: Feasibility of Remote Cochlear Implant Users' Follow-up
Acronym: TELERIC1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital Rothschild (Other)
Responsible Party: Principal Investigator, Christine PONCET-WALLET, head of Service CRIC ENT Hôpital Rothschild, Hôpital Rothschild
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 2014-A01871-46
Record Dates: First submitted 2017-01-12; First posted 2017-01-16 (Estimated); Last update posted 2017-10-02 (Actual); Status verified 2017-01

CONDITIONS: Deafness; Perception, Bilateral
Keywords: cochlear implant ;
MeSH Terms: conditions — Deafness | interventions — Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- group A start with the remote session followed by on site (Experimental)
  Interventions: Other: telemedicine
- group B start with on site followed by telemedecine (Active Comparator)
  Interventions: Other: telemedicine

INTERVENTIONS:
Other: telemedicine — telemedicine applied to adult cochlear implant users' follow-up

SUMMARY:
Cochlear implants (CIs) are medical devices now widely used in persons with severe to profound hearing loss. After a six month to one-year period following implantation, adults typically reach optimal fitting parameters, which lead to a stabilized hearing performance with their CI. At this stage, they usually enter a routine clinical after-care program, which involves regular appointmentsattheir CI center. Such visits aim at identifying any complication, which can be medical (abnormal cutaneous healing evolution) and/or device related, as well as any declinein performance (possibly related to the former). In France, the HAS (French Health Authority) recommends CI users tobe seen around threetimes a year during the second and third years after implantation, and then annually. While the schedule of appointments remains dependent on centers' practices, there is some kind of consensus about the minimal content of a long-term follow-up session:medical consultation, CI external parts checking, free field aided tonal audiometry, fitting adjustments if necessary,speech understanding assessments.

Our center (CRIC) is one of the biggest French CI implant centers approved by the HAS, providing after-care for no less than 750 CI users, most of whomhave entered their long-term follow-up period. For some, attending follow-up appointments may need several hours, require taking a half-day off work, and entail travel expenses. Some patients may also have associated disabilities making it difficultto reach the center.Moreover, although the cohort of patients has increased over the years, the number of trained professionals and the clinical care infrastructures have not evolved proportionally. As a consequence, there is a need to reduce the number of routine visits, to allow more scope for complex cases andto efficiently identify issues.

Remote consultation seems to address all the points listed above. However, it appears that little has been doneto develop remote after-care for cochlear implant recipients. Published studies mainly focus on the fitting aspects.

The development of telemedicine has become one of the key priorities of the French government over the past few years, and it is now feasible thanks to the development of high speed connections (ADSL, mobile internet, high definition transmissions). Promoting telemedicine has several goals, the main one being to extend health care services to underserved patients in remote locations; it also allows some medical units to be freed upand to reserve infrastructures and professionals for patients requesting critical care. Of course, telemedicine is also meant to save costs.

The objectif of this protocole is to evaluate the feasibility of telemedicine applied to adult cochlear implant users' follow-up by comparing the data of the medical consultation and speech therapy assessment, carried out in the CRIC service and videoconferencing when the patient is home, using his computer equipment to communicate with the CRIC.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cochlear implants for more than 12 months followed by CRIC
* native French language
* possibility to carry out the sessions (remote and on-site) within a short time (30 days +/- 8 days) .Patients who can have a computer with internet connection quality and user of remote access type Skype in good conditions Listening, privacy and anonymity.
* Having given their consent to participate in this protocol

Exclusion Criteria:

* Unavailability to carry out the acts of telemedicine
* Difficulty having good quality remote access from home
* Not benefiting from a social protection scheme
* Persons deprived of their liberty by judicial or administrative decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
comparison the data of the medical consultation and speech therapy assessment, carried out in the CRIC service and videoconferencing when the patient is home, using his computer equipment to communicate with the CRIC | 18 months
  No differences between the speech data and the consultation data for acts at a distance compared to face-to-face acts.

IPD SHARING:
Plan to Share IPD: No